CLINICAL TRIAL: NCT03818906
Title: Efficacy of aPDT in Reducing Pain and Swelling Following Molar Extraction Surgery- Blinded Randomized Controlled Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Principal Investigator, Livia Azeredo Alves Antunes, Professor Lívia Azeredo Alves Antunes, Universidade Federal Fluminense
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PDTa and reducing pain
Record Dates: First submitted 2019-01-24; First posted 2019-01-28 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Tooth Extraction Status Nos
Keywords: Photochemotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Group (Active Comparator): Patients with first or second molars where the extractions will be performed in a conventional way without any additional local treatment to be done in the alveolus. The analysis of the postoperative signs/symptoms will be performed by the visual analog pain scale at 1th, 2th, 3th, 4th, 5th, 6th, 7th. Subjective evaluation of swelling in 48 hours and 7th day.
  Interventions: Procedure: Molar extraction - Control Group
- Test Group 1 (Experimental): Patients with first or second molars where the extractions will be performed in a conventional way and after extraction will be performed aPDT inside the alveolus.The analysis of the postoperative signs/symptoms will be performed by the visual analog pain scale at 1th, 2th, 3th, 4th, 5th, 6th, 7th. Subjective evaluation of swelling in 48 hours and 7th day.
  Interventions: Procedure: aPDT + Molar Extraction - Test Group 1
- Test Group 2 (Experimental): Patients with first or second molars where the extractions will be performed in a conventional way and immediately after the exodontia, the fresh socket will receive local application of infrared in the outer vestibular portion. The analysis of the postoperative signs/symptoms will be performed by the visual analog pain scale at 1th, 2th, 3th, 4th, 5th, 6th, 7th. Subjective evaluation of swelling in 48 hours and 7th day.
  Interventions: Procedure: Infrared + Molar Extraction - Test Group 2
- Test Group 3 (Experimental): Patients with first or second molars where the extractions will be performed in a conventional way and immediately after the exodontia the approaches from the previous groups (Test Group 1 and 2 (aPDT + infrared) will be done. The analysis of the postoperative signs/symptoms will be performed by the visual analog pain scale at 1th, 2th, 3th, 4th, 5th, 6th, 7th. Subjective evaluation of swelling in 48 hours and 7th day.
  Interventions: Procedure: aPDT + Infrared + Molar Extraction - Test Group 3

INTERVENTIONS:
Procedure: Molar extraction - Control Group — The extra-oral measurements will be made for further comparison and assessment of swelling (48 hours and 7 days). Exodontia will be done in a conventional way and the evolution of the pain will be evaluated through the visual analog scale during the next 7 days.
  Arms: Control Group
Procedure: aPDT + Molar Extraction - Test Group 1 — The extra-oral measurements will be made for further comparison and assessment of swelling (48 hours and 7 days). Exodontia will be done in a conventional way and the evolution of the pain will be evaluated through the visual analog scale during the next 7 days.immediately after extraction, the fresh sockets will receive in their internal portion a local application of aPDT.
  Arms: Test Group 1
Procedure: Infrared + Molar Extraction - Test Group 2 — The extra-oral measurements will be made for further comparison and assessment of swelling (48 hours and 7 days). Exodontia will be done in a conventional way and the evolution of the pain will be evaluated through the visual analog scale during the next 7 days.immediately after extraction, the fresh sockets will receive local application of infrared in vestibular external portion
  Arms: Test Group 2
Procedure: aPDT + Infrared + Molar Extraction - Test Group 3 — The extra-oral measurements will be made for further comparison and assessment of swelling (48 hours and 7 days). Exodontia will be done in a conventional way and the evolution of the pain will be evaluated through the visual analog scale during the next 7 days.immediately after extraction, the fresh sockets will receive in their internal portion a local application of aPDT and after that will receive local application of infrared in vestibular external portion.
  Arms: Test Group 3

SUMMARY:
This project aims to evaluate the effect of antimicrobial photodynamic therapy (aPDT) on the reduction of swelling and postoperative pain in lower molar extraction procedures. This is a clinical study approved by the Research Ethics Committee, which will be performed in 40 patients between 20 and 60 years. Patients included in the study should have at least one lower molar (first or second molar) with indication of exodontia. Participants will follow the exclusion criteria: pregnant or breastfeeding women; patients with obesity (Body Mass Index - BMI); make use of any activity smokers and ex smoker to 6 months; diabetics; immunosuppressed; in osteoporosis; making use of antimicrobials in the last 3 months; making use of medications that interfere with bone remodeling; with cysts or tumors in place. Surgical procedures that exceeded the clinical time of 30 minutes and / or required opening of the flap or osteotomy were excluded from the study. After the sample calculation, forty patients will be involved in this project, where forty molars (first and second molars) will be extracted in the mandible, which will be randomly divided into 4 groups. The control group (C.G), will contain 10 patients, where 10 molars will be extracted in a conventional way, without any additional treatment to be done. Test group 1 (T.G1) will contain 10 patients where 10 molars will be extracted and immediately after extraction, the fresh sockets will receive in their inner portion a local application of aPDT. The test group 2 (T.G2) will present 10 patients, where 10 molars will be extracted that immediately after the exodontia, the fresh socket will receive local application of infrared in the outer vestibular portion. Finally, Test Group 3 (T.G3), will be composed of 10 patients, where 10 molars will be extracted, joining the approaches of the previous groups (aPDT + infrared). Pain intensity will be assessed through a visual analogue scale and swelling assessed by measuring a perimeter between the tragus, the base of the jaw and the commissure of the lips. The data will be collected in four moments: before the surgery, 72 hours, 7 days and 30 days postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* patients without systemic limitations that indicate surgical procedures with cooperative behavior
* with full awareness and approval of the guidelines listed in the free and clarified term proposed by the research
* present compromised posterior and inferior teeth requiring exodontia.

Exclusion Criteria:

* Pregnant or breastfeeding women
* Patients with obesity (Body Mass Index - BMI)
* Make use of any activity smokers and ex smoker to 6 months
* Diabetics
* Immunosuppressed
* in osteoporosis
* making use of antimicrobials in the last 3 months
* making use of medications that interfere with bone remodeling
* with cysts or tumors in place
* Surgical procedures that exceeded the clinical time of 30 minutes and / or required opening of the flap or osteotomy

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
reduction of postoperative pain | Pain evaluation will be performed prior to the surgical procedure and 7 days after
  Evaluate Antimicrobial photodynamic therapy (aPDT)on the reduction of postoperative pain in lower molar extraction procedures. Pain intensity will be assessed through a visual analogue scale
reduction of swelling | The data will be collected in four moments: before the surgery, 72 hours, 7 days and 30 days postoperatively.
  Evaluate Antimicrobial photodynamic therapy (aPDT)on the reduction of swelling. Swelling evaluated through the measurement of a perimeter between the tragus, the base of the mandible and the commissure of the lips

CONTACTS AND LOCATIONS:
Locations (1):
- Livia Antunes, PhD, Nova Friburgo, Rio de Janeiro, Brazil